CLINICAL TRIAL: NCT06775080
Title: The Use of Propranolol in the Perioperative Period of Resectable Gastrointestinal Tumors and the Study of Its Immune Mechanism Research
Brief Title: The Use of Propranolol in the Perioperative Period of Resectable Gastrointestinal Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhongguang Luo, MD, Chief Physician, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1317
Record Dates: First submitted 2024-12-27; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- propranolol (beta-blocker used treat high blood pressure)+surgeries (Experimental)
  Interventions: Drug: propranolol (beta-blocker used treat high blood pressure)

INTERVENTIONS:
Drug: propranolol (beta-blocker used treat high blood pressure) — Enrolled patients began receiving propranolol alone orally twice daily (10 mg bid) 10-14 days prior to surgery, and after 3 days of treatment, the dose of propranolol was increased to 20 mg bid daily until the day of surgery if the following three predefined criteria were met: systolic blood pressure greater than 90 mmHg, heart rate greater than 60 bpm, and no significant symptoms (e.g., syncope, insomnia, fatigue). The patient continues to be treated from 1 week after surgery.From 1 week after surgery, patients continue propranolol for 3 weeks. Patients will be monitored daily for symptoms, blood pressure, and heart rate and will be followed for observation at 6, 12, and 24 months after surgery until disease progression or clinical death, unless intolerable toxicity occurs and the patient refuses to continue treatment. The efficacy and safety of the preoperative propranolol β-blockade regimen in patients with gastrointestinal tract tumors was evaluated using the study objectives in S

SUMMARY:
In this study, perioperative propranolol β-blockade was administered to patients with surgically resectable primary gastrointestinal tumors to explore the safety, efficacy, and alleviation of perioperative psychological stress. At the same time, a multi-omics study was conducted using clinical samples to explore the activation of anti-tumor immune response and its mechanism.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled pilot exploratory clinical study to enroll 20 patients with surgically resectable primary gastric cancer and 20 patients with surgically resectable primary colorectal cancer. Each enrolled patient will be assigned a case number. This case number and the patient's initials will be entered on each page of the case report form. Trial group (10 patients with gastric cancer and 10 patients with intestinal cancer): Enrolled patients will be hospitalized for 10-14 days of preoperative propranolol β-blockade monotherapy prior to surgery (including the day of surgery) for evaluation of efficacy and safety. Control group (10 cases of gastric cancer and 10 cases of intestinal cancer): no propranolol drug treatment. Patients will be observed during the treatment period and at 6 months, 12 months and 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Surgically resectable primary gastric cancer and colorectal cancer;
2. Age greater than 18 years old and less than 65 years old;
3. Negative pregnancy test for women of childbearing age;
4. ECOG score ≤2;
5. Signed informed consent.
6. Resting blood pressure greater than 100/60mmHg, heart rate greater than 60 beats per minute.

Exclusion Criteria：

1) Pregnant or breastfeeding women, or women with pregnancy plans within six months; 2) Patients with absolute or relative contraindications to propranolol:

1. Pathological sinus node syndrome;
2. Sinus bradycardia (less than 60 beats/minute);
3. First, second or third degree AV block;
4. Resting blood pressure less than 100/60 mmHg;
5. untreated pheochromocytoma;
6. untreated thyroid disease;
7. Patients on dihydropyridine or non-dihydropyridine calcium channel blockers (e.g., diltiazem, verapamil, nifedipine, amlodipine);
8. Severe peripheral vascular disease (intermittent claudication);
9. Patients on antiarrhythmic drugs (e.g., amiodarone, sotalol, digoxin);
10. Patients with renal insufficiency (defined as creatinine clearance greater than 0.15 mmol/L);
11. Patients with hepatic insufficiency: AST or ALT or ALP > 2.5 times the upper limit of normal (ULN), bilirubin > 1.5 times the ULN, ALP > 2.5
12. Patients using colistin, digoxin, rizatriptan, cimetidine, hydralazine, guanethidine, or ergotamine.
13. Patients with a history of major depressive episodes; 3) Patients who have undergone surgery for GI tumors within the previous six months; 4) Patients receiving neoadjuvant chemotherapy prior to planned gastrointestinal tumor resection; 5) patients using conventional anxiolytic drugs (e.g. benzodiazepines), alpha-adrenergic agonists (e.g. colistin); 6) Patients using selective or non-selective β-adrenergic inhibitors (e.g., propranolol, metoprolol, atenolol, sotalol) within the last three months; 7) Patients with a history of stroke; 8) Patients with moderate or severe asthma, defined as requiring hospitalization or oral steroid therapy; (9) Those who, in the opinion of the physician, have other reasons for not being included in the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Depression Scale Scores | Within two years of enrollment
  Hamilton Anxiety Scale. The higher the score, the worse the symptoms.
heart rate | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
Heart rate variability | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
blood preasure | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
Norepinephrine levels | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
blood glucose | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
SaO2 | From enrollment to 24 days postoperatively
  Sympathetic nervous system activation index
RNA-seq of tumor tissue | Baseline and during surgery
  Tumor tissues were examined by RNA-seq to assess the alteration of tumor microenvironment before and after treatment, and to explore the possible alteration of activation pathways (DAMP, RIG-I, NF-kB, JAK-STAT, etc.).
RNA-seq of peripheral blood PBMCs | Baseline and during surgery
  Peripheral blood PBMCs were examined by RNA-seq to assess the alteration of tumor microenvironment before and after treatment, and to explore the possible alteration of activation pathways (DAMP, RIG-I, NF-kB, JAK-STAT, etc.).
Flow cytometry of peripheral blood PBMC | Baseline and during surgery
  Flow cytometry was applied to the peripheral blood PBMC to assess the changes in the systemic immune system and tumor immune microenvironment before and after treatment, and to explore new subpopulations of immune cells with characteristic alterations.
Flow cytometry of tumor tissues | Baseline and during surgery
  Flow cytometry was applied to the tumor tissues to assess the changes in the systemic immune system and tumor immune microenvironment before and after treatment, and to explore new subpopulations of immune cells with characteristic alterations.
ELISA detection of tumor tissue | Baseline and during surgery
  Tumor tissues were examined using ELISA to explore functional changes in specific immune cell subsets before and after preoperative propranolol treatment.
ELISA detection of peripheral blood PBMCs | Baseline and during surgery
  Functional changes in specific immune cell subsets before and after preoperative propranolol treatment were explored using ELISA for peripheral blood PBMC.

SECONDARY OUTCOMES:
2-year OS rate | Two years after surgery
2-year RFS rate | Two years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China